CLINICAL TRIAL: NCT03323788
Title: PGC-1 & MUSCLE MITOCHONDRIAL DYSFUNCTION IN DIABETES: AIMS 1-4
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Lawrence Mandarino, Professor of Medicine, University of Arizona
Other Study IDs: 1606632517
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Type2 Diabetes; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Aim 1: Aim 1. To determine whether the transcription factor expression response to exercise is dysregulated in muscle from type 2 diabetic patients. We will test the hypothesis that MZF1, NFKB1, RELA, SP1/KLF and EGR1 responses to an acute exercise bout are reduced in insulin resistant patients with type 2 diabetes.
- Aim 2: Aim 2. To determine how insulin resistance changes the response of post-translational modifications of SP1/KLF family and MZF1 transcription factors to acute exercise in muscle from type 2 diabetic patients. We will test the hypothesis that:
  1. SP1/KLF2, 4, and 6 and phosphorylation/acetylation and MZF1 phosphorylation is altered in response to acute exercise.
  2. The response of SP1/KLF2, 4, and 6 phosphorylation and acetylation and MZF1 phosphorylation to acute exercise is abnormal in patients with type 2 diabetes.
- Aim 3: Aim 3. To define the response of miRNAs to acute exercise in healthy and insulin resistant muscle from obese and type 2 diabetic patients. We will test the hypotheses that:
  1. The exercise-induced increases in expression of miR-378 members and miR-128 are lower in obese and type 2 diabetic muscle than in lean healthy controls.
  2. FOXO1 expression, a target of miR-378 and miR-128, is higher in obese and type 2 diabetic muscle and this is accompanied by decreased FOXO1 phosphorylation.
  3. The exercise-induced increases in expression of miR-30 family members, miR-10a, miR-422a, and miR-532 are lower in obese and type 2 diabetic muscle.
  4. There are novel miRNAs that regulate the transcriptional program induced by acute exercise and are dysregulated in insulin resistance.
- Aim 4: Aim 4. To determine whether treatment with PPAR-Alpha agonist fibrate derivatives suppresses the normal gene expression response to acute exercise. We will test the hypothesis that Gemfibrozil treatment inhibits the normal transcriptional response to exercise.

SUMMARY:
We are trying to understand how insulin (a type of hormone in the body that regulates how the body regulates how one metabolizes protein and carbohydrates) and exercise alter proteins involved in energy production and metabolism in skeletal muscle.

DETAILED DESCRIPTION:
(Aims 1-3) We are trying to understand how insulin (a type of hormone in the body that regulates how the body regulates how one metabolizes protein and carbohydrates) and exercise alter proteins involved in energy production and metabolism in skeletal muscle. By studying this, they hope to better understand the causes of insulin resistance and Type 2 diabetes Insulin is a hormone that is produced normally in the body and causes blood sugar to return to normal after eating. Insulin resistance is a state when the body is not using insulin correctly, and more insulin is needed to keep blood sugar concentrations normal. Insulin resistance can lead to Type 2 diabetes. Type 2 diabetes is a disease in which blood sugar levels are too high. Our studies may help to find out why some people develop Type 2 diabetes and how exercise may prevent this disease.

(Aim 4) We are asking patients from aims 1-3 to take part in this research study because they have high triglycerides that could be treated anyway with fibrates, and they do not have diabetes.

Triglycerides and cholesterol are the two main kinds of fat that are in blood. People who have high triglycerides have some health risks and are sometimes treated with drugs called "fibrates". This drug turns on a protein in ones body that controls the activity of some of the genes that make it easier for their liver to get rid of triglycerides. We think that maybe this same gene, in ones muscle, can lower the ability of genes in ones muscle to respond beneficially to exercise, but we don't know if this is true.

ELIGIBILITY:
Aims 1-3.

1. Age 30-59
2. BMI: Lean, BMI less than or equal to 25; Obese, BMI between 30- 50; type 2 diabetic, BMI between 30- 50.
3. Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
4. Subjects may be of either sex with age as described in each protocol. Female subjects must be non-lactating and will be eligible only if they have a negative pregnancy test throughout the study period.
5. Subjects must range in age as described in each specific protocol.
6. Subjects must have the following laboratory values:

   1. Hematocrit ≥ 35 vol%
   2. Serum creatinine ≤ 1.6 mg/dl
   3. AST (SGOT) < 2 times upper limit of normal
   4. ALT (SGPT) < 2 times upper limit of normal
   5. Alkaline phosphatase < 2 times upper limit of normal
   6. Triglycerides < 150 mg/dl for nondiabetics (except for Aim 4).
   7. Triglycerides <300 for diabetics (except for Aim 4)
   8. INR ≤ 1.3 Aim 4

1. Age 30-59 2. BMI: Lean, BMI less than or equal to 25; Obese, BMI between 30- 50. 3. Patients may have normal or impaired glucose tolerance. 4. Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.

5. Subjects may be of either sex with age as described in each protocol. Female subjects must be non-lactating and will be eligible only if they have a negative pregnancy test throughout the study period.

6. Subjects must have the following laboratory values:

1. Hematocrit ≥ 35 vol%
2. Serum creatinine ≤ 1.6 mg/dl
3. AST (SGOT) < 2 times upper limit of normal
4. ALT (SGPT) < 2 times upper limit of normal
5. Alkaline phosphatase < 2 times upper limit of normal
6. Triglycerides > 300 mg/dl for nondiabetics, > 250 mg/dl for impaired glucose tolerance.
7. INR ≤ 1.3 7. Patients must be prescribed gemfibrozil from their doctor

Exclusion Criteria:

* 1. Subjects must not be receiving any of the following medications: thiazide or furosemide diuretics, beta-blockers, or other chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on a stable dose of such agents for the past three months before entry into the study. Subjects may be taking a stable dose of estrogens or other hormonal replacement therapy, if the subject has been on these agents for the prior three months. Subjects taking systemic glucocorticoids are excluded. Patients with type 2 diabetes will be excluded if they are taking thiazolidinediones, but may be taking sulfonylureas or other medications known to work through effects on insulin sectretion.

  2. Subjects receiving Gemfibrozil must not also be receiving a statin. 3. Subjects with a history of clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.

  4. Recent systemic or pulmonary embolus, untreated high-risk proliferative retinopathy, recent retinal hemorrhage, uncontrolled hypertension, systolic BP>180, diastolic BP>105, autonomic neuropathy, resting heart rate >100, electrolyte abnormalities.

Ages: 30 Years to 59 Years | Sex: All
Age Groups: Adult
Study Population: The plan is to have about 84 people take part in aims 1 to 3 and about 12 people in aim 4. Adults between the ages of 30 - 59 may participate.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Response of muscle mRNA to acute exercise | 2014-2019
  mRNA differential response in muscle to exercise in obese patients

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Mandarino, PHD, Principal Investigator — The University of Arizona
Locations (1):
- The University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No